CLINICAL TRIAL: NCT06122298
Title: Testing the Interplay of Gambling, Emotion and Reward
Acronym: TIGER
Status: Recruiting | Type: Observational
Sponsor: Hôpital le Vinatier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-A00597-38
Record Dates: First submitted 2023-09-28; First posted 2023-11-08 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Gambling Addiction
Keywords: gambling addiction; fMRI; reward; emotion; striatum; amygdala; EMA
MeSH Terms: conditions — Gambling | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with gambling problems: This group includes individuals suffering from gambling addiction as defined by the DSM-5, and individuals suffering from "problem gambling", just below the DSM-5 diagnostic threshold.
  Interventions: Other: fMRI; Other: Ecological Momentary Assessment
- Healthy control individuals: Matched healthy individuals
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — A brain imaging technique that measures in vivo the activity of brain areas by detecting local changes in blood flow.
Other: Ecological Momentary Assessment — studies people's thoughts and behaviour in their daily lives by repeatedly collecting data in an individual's normal environment, at or close to the time they carry out that behaviour
  Other Names: EMA
  Groups: Individuals with gambling problems

SUMMARY:
Background The nature and direction of dysfunctional reward processing in gambling disorder remains unclear. We aim to test a novel neurobiological model of gambling addiction, that takes into account inter-individual differences, as well as the multifactorial nature of gaming addiction.

Objectives

Primary objective:

This project will test the hypothesis that there are two opposite brain phenotypes that characterize two distinct subpopulations of gamblers, so-called impulsive vs. emotional, respectively.

Secondary objective:

This project will also seek to determine whether the brain phenotypes proposed above are capable of predicting gambling behavior outside the laboratory.

Study design The primary objective will be tested using a reward task and a facial emotion recognition task performed by participants in an fMRI scanner.

The secondary objective will be tested by combining fMRI measures with behavioral measures from everyday life collected via Ecological Momentary Assessment (EMA).

Study population This study will focus on individuals with gambling problems, as well healthy subjects with no gambling problems and no psychiatric comorbidities.

Outcomes/Endpoints

Primary endpoint:

We will compare striatum and amygdala reactivity between the three groups of impulsive gamblers, emotional gamblers and healthy subjects.

Secondary endpoint:

We will assess the correlation between emotional states and gambling behavior in everyday life, based on striatum and amygdala reactivity, using multiple linear regression models.

DETAILED DESCRIPTION:
Background Gambling addiction has often been conceptualized as the result of reward processing dysfunction in the brain, particularly in the striatum, a key structure of the reward system. Although a number of studies have provided support for this hypothesis, neuroimaging studies have produced inconsistent results, suggesting either hypo- or hyper-reactivity to rewards in gambling addiction. These inconsistencies have been the subject of intense debate, but remain unexplained to this day, hampering our understanding of the disease and the development of effective therapeutic strategies. The aim of this project is to test a new neurobiological model of gambling addiction that has the potential to reconcile these inconsistencies. A particular feature of this model is that it takes into account inter-individual differences, as well as the multifactorial nature of gaming addiction.

Objectives

Primary objective:

This project will test the hypothesis that there are two opposite brain phenotypes in gambling addiction: striatal hyper-reactivity to reward combined with amygdala hypo-reactivity to emotional stimuli, and striatal hypo-reactivity to reward combined with amygdala hyper-reactivity to emotional stimuli. The investigators further hypothesize that these two brain phenotypes characterize two distinct subpopulations of gamblers, so-called impulsive vs. emotional, respectively.

Secondary objective:

This project will also seek to determine whether the brain phenotypes proposed above are capable of predicting gambling behavior outside the laboratory. To do this, the investigators will use Ecological Momentary Assessment (EMA), which involves using participants' smartphones to perform repeated, real-time sampling of their gambling behavior and emotions in real life. The investigators hypothesize that a significant difference in reactivity between the striatum and the amygdala will be associated with a strong correlation between 1) gambling behavior and positive emotions in impulsive gamblers, and 2) gambling behavior and negative emotions in emotional gamblers.

Study design The primary hypothesis will be tested using cognitive tasks performed by participants in an fMRI scanner. In order to assess striatal reactivity to reward, the investigators will use fMRI combined with a reward task. The investigators will use fMRI combined with a facial emotion recognition task to measure the reactivity of the amygdala to emotional stimuli. These tasks will allow the investigators to establish the brain phenotypes characterizing impulsive and emotional gamblers, and test the hypothesis that these phenotypes are diametrically opposed in these two sub-populations.

The secondary hypothesis will be tested by combining fMRI measures with behavioral measures from everyday life (EMA). In concrete terms, gamblers will be followed longitudinally for up to 4 weeks, and will receive short questionnaires 3 to 4 times a day on their smartphones to assess their gambling behavior (number of hours spent gambling, amount of money spent...) as well as their emotions (positive and negative). These measurements will enable the investigators to test the hypothesis that the brain phenotypes described above are capable of predicting the relationship between emotions and gambling behavior in everyday life.

Study population This study will focus on individuals with gambling problems. This category includes individuals suffering from gambling addiction as defined by the DSM-5, and individuals suffering from "problem gambling", just below the DSM-5 diagnostic threshold. Extending recruitment to individuals with problem gambling should facilitate recruitment, while considering the existence of a continuum of gambling problems.

The study will also include a control group of healthy subjects with no gambling problems and no psychiatric comorbidities.

The plan is to recruit 60 gamblers and 60 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

For all participants (gamblers and healthy subjects)

* Aged between 18 and 65
* Fluent French, read and spoken
* Male and Female
* Informed consent to take part in the research

For gamblers :

* Number of DSM-5 critera for gambling disorder ≥3
* Score ≥ 5 on the Problem Gambling Severity Index questionnaire (PGSI)
* Have a smartphone

For healthy subjects :

* no DSM-5 criteria for gambling addiction
* Score ≤ 2 on the Problem Gambling Severity Index questionnaire (PGSI)

Exclusion Criteria:

For all participants (gamblers and healthy subjects):

* Contra-indication to MRI
* Protected Adults
* Breast feeding or pregnant women
* Neurological disorder or severe chronic illness (diabetes, heart disease, kidney disease, lung disease or liver disease, inflammatory disease….)
* Pharmacological treatment with psychotropic action (>1 time / week)
* Regular drug use (> 1 time/ week for at least 3 months in the last 6 months)
* Positive urine drug test on the day of the MRI sessions

For gamblers:

* Psychiatric treatment > 1 month (pharmacological or CBT)
* Other DSM-5 diagnosis : schizophrenia, bipolar disorder, ADHD, autism, current PTSD, eating disorders, current major depressive episode, anxiety disorder, substance use disorder except nicotine, obsessive compulsive disorder.

For healthy subjects :

- Any DSM-5 diagnosis except nicotine addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups: 60 individuals with gambling problems (i.e. Number of DSM-5 critera for gambling disorder ≥3) and 60 matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Striatal BOLD response to reward outcomes and amygdala BOLD response to emotional stimuli | 4 weeks
  Striatal BOLD response: average BOLD signal as measured with fMRI in the striatum in response to monetary reward outcomes in a gambling task.
  amygdala BOLD response: average BOLD signal as measured with fMRI in the amygdala in response to emotional faces in a facial emotion recognition task.

SECONDARY OUTCOMES:
Correlation between emotional states and gambling behavior in everyday life | 4 weeks
  Emotions and gambling behavior in everyday life will be measured using Ecological Momentary Assessment on gamblers' smartphones

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume SESCOUSSE, PHD, Principal Investigator — CH Le Vinatier
Locations (1):
- CH le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No